CLINICAL TRIAL: NCT02250248
Title: AttraX® Putty vs. Autograft in eXtreme Lateral Interbody Fusion (XLIF®): A Prospective Randomized Single-Center Evaluation of Radiographic and Clinical Outcomes
Brief Title: AttraX® Putty vs. Autograft in XLIF®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NUVA.AX1401
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Conditions of the Lumbar Spine
Keywords: Degenerative disc disease; Lumbar spine
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AttraX Putty (Active Comparator): Patient will be treated with AttraX Putty intraoperatively.
  Interventions: Biological: AttraX Putty
- Iliac Crest Bone Graft (ICBG) (Active Comparator): Patients will be treated with ICBG harvested during surgery.
  Interventions: Other: Iliac Crest Bone Graft (ICBG)

INTERVENTIONS:
Biological: AttraX Putty
  Arms: AttraX Putty
Other: Iliac Crest Bone Graft (ICBG)
  Other Names: autograft
  Arms: Iliac Crest Bone Graft (ICBG)

SUMMARY:
The objective of this study is to evaluate the clinical success of AttraX Putty as a bone graft substitute for autograft in XLIF procedures.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized study. Subjects will be recruited from patients already under the Investigator's care who are indicated for XLIF with iliac crest bone graft (ICBG) autograft or AttraX Putty. To minimize bias, all consecutive patients at a given investigational site who meet eligibility requirements will be asked to consent to participate in the study whereby the biologic (ICBG autograft or AttraX Putty) will be randomly assigned. All subjects will be followed for 24 months following surgery to quantify the clinical and radiographic improvements of each biologic compared to baseline and in comparison with each other.

ELIGIBILITY:
Inclusion Criteria:

1. Persistent back and/or leg pain unresponsive to conservative treatment for at least 6 months, unless surgical treatment is clinically indicated sooner
2. Indicated for a single-level XLIF between L1 and L5 with bilateral percutaneous pedicle screws
3. Objective evidence of primary diagnosis must be confirmed by appropriate imaging studies
4. 18-80 years of age at the date of written informed consent
5. Able to undergo surgery based on physical exam, medical history, and surgeon judgment
6. Expected to survive at least 2 years beyond surgery
7. Willing and able to return for post-treatment exams according to the follow-up called for in the protocol
8. Signed and dated informed consent form

Exclusion Criteria:

1. Mental or physical condition that would limit the ability to comply with study requirements
2. Spine abnormality requiring treatment at more than one level
3. Previous failed fusion at any spinal level
4. Prior fusion procedure at operative level (i.e., no revision of operative level)
5. Prior adjacent level fusion (note: prior decompression is not an exclusion)
6. Systemic or local infection; active or latent
7. Diseases that significantly inhibit bone healing (e.g., prior diagnosis of osteoporosis, metabolic bone disease)
8. Treatment with pharmaceuticals interfering with calcium metabolism
9. Undergoing chemotherapy or radiation treatment
10. Chronic use of steroids (defined as more than 6 weeks of steroid use within 12 months of surgery, other than episodic use or inhaled corticosteroids)
11. Involvement in active litigation relating to the spine (worker's compensation claim is allowed if it is not contested)
12. Significant general illness (e.g., HIV, active metastatic cancer of any type, uncontrolled diabetes, dialysis dependent renal failure, symptomatic liver disease)
13. Immunocompromised or is being treated with immunosuppressive agents
14. Pregnant, or plans to become pregnant during the study
15. Subject is a prisoner
16. Participating in another clinical study that would confound study data
17. At risk to be non-compliant (e.g. (recently treated for) substance abuse, detainee, likely to immigrate)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
The number and percentage of subjects with radiographically apparent fusion 24 months. | 24-months
  The number and percentage of subjects with radiographically apparent fusion 24 months.

SECONDARY OUTCOMES:
The rate of complications attributable to the use of AttraX and ICBG autograft. | Post-op to 24-months
  The rate of complications attributable to the use of AttraX and ICBG autograft.
The change in self-reported clinical outcomes scores from baseline through 24 month follow-up, including VAS (back, leg, and iliac crest pain), ODI, EQ5D, and SF-36. | Pre-op through 24-months
  The change in self-reported clinical outcomes scores from baseline through 24 month follow-up, including VAS (back, leg, and iliac crest pain), ODI, EQ5D, and SF-36.
The morbidity associated graft harvest as measured by operative time, blood loss, length of hospital stay, postoperative pain, and infection rate. | Surgery through 24-months
  The morbidity associated graft harvest as measured by operative time, blood loss, length of hospital stay, postoperative pain, and infection rate.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano M Menezes, M.D., Principal Investigator — Lifecenter to Mater Dei Hospital
Locations (1):
- Mater Dei Hospital, Barro Prêto, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No